CLINICAL TRIAL: NCT00493220
Title: INcreased Flow Utilizing Subcutaneously-Enabled Ceftriaxone (INFUSE-Ceftriaxone) Study: A Phase I Study Comparing the Safety and Pharmacokinetics of Ceftriaxone Administered Subcutaneously With and Without Human Recombinant Hyaluronidase (HYLENEX Recombinant) and Intravenously in Human Volunteers
Brief Title: Pharmacokinetic and Safety Study of HYLENEX Recombinant-Augmented Subcutaneous Ceftriaxone Administration
Acronym: INFUSE-Cftrx
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Collaborators: Halozyme Therapeutics (Industry)
Responsible Party: Geroge E. Harb, MD, Baxter Healthcare Corporation
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1838-004
Record Dates: First submitted 2007-06-26; First posted 2007-06-28 (Estimated); Results first posted 2011-12-02 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-10

CONDITIONS: Healthy
Keywords: ceftriaxone; cephalosporins; pharmacokinetics; subcutaneous; hyaluronoglucosaminidase; hyaluronidase; hyaluronan; rHuPH20
MeSH Terms: interventions — Ceftriaxone; Hyaluronoglucosaminidase; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- HYLENEX SC, Placebo SC, IV (Experimental): subcutaneous HYLENEX and ceftriaxone as 1st intervention, subcutaneous placebo and ceftriaxone as 2nd intervention, IV ceftriaxone as 3rd intervention
  Interventions: Drug: SC HYLENEX and Ceftriaxone; Drug: SC Placebo and Ceftriaxone; Drug: IV Ceftriaxone
- HYLENEX SC, IV, Placebo SC (Experimental): subcutaneous HYLENEX and ceftriaxone as 1st intervention, IV ceftriaxone as 2nd intervention, subcutaneous placebo and ceftriaxone as 3rd intervention
  Interventions: Drug: SC HYLENEX and Ceftriaxone; Drug: SC Placebo and Ceftriaxone; Drug: IV Ceftriaxone
- Placebo SC, HYLENEX SC, IV (Experimental): subcutaneous placebo and ceftriaxone as 1st intervention, subcutaneous HYLENEX and ceftriaxone as 2nd intervention, IV ceftriaxone as 3rd intervention
  Interventions: Drug: SC HYLENEX and Ceftriaxone; Drug: SC Placebo and Ceftriaxone; Drug: IV Ceftriaxone
- Placebo SC, IV, HYLENEX SC (Experimental): subcutaneous placebo and ceftriaxone as 1st intervention, IV ceftriaxone as 2nd intervention, subcutaneous HYLENEX and ceftriaxone as 3rd intervention
  Interventions: Drug: SC HYLENEX and Ceftriaxone; Drug: SC Placebo and Ceftriaxone; Drug: IV Ceftriaxone
- IV, HYLENEX SC, Placebo SC (Experimental): IV ceftriaxone as 1st intervention, subcutaneous HYLENEX and ceftriaxone as 2nd intervention, subcutaneous placebo and ceftriaxone as 3rd intervention
  Interventions: Drug: SC HYLENEX and Ceftriaxone; Drug: SC Placebo and Ceftriaxone; Drug: IV Ceftriaxone
- IV, Placebo SC, HYLENEX SC (Experimental): IV ceftriaxone as 1st intervention, subcutaneous placebo and ceftriaxone as 2nd intervention, subcutaneous HYLENEX and ceftriaxone as 3rd intervention
  Interventions: Drug: SC HYLENEX and Ceftriaxone; Drug: SC Placebo and Ceftriaxone; Drug: IV Ceftriaxone

INTERVENTIONS:
Drug: SC HYLENEX and Ceftriaxone — single, subcutaneous, 150 U dose of HYLENEX; followed by single, subcutaneous, 1 gm dose of ceftriaxone (350 mg/mL solution administered at 2.5 mL/min over 1.14 minutes)
  Other Names: HYLENEX recombinant; hyaluronoglucosaminidase; hyaluronidase; rHuPH20
Drug: SC Placebo and Ceftriaxone — single, subcutaneous injection of 1 mL 0.9% sodium chloride solution; followed by single, subcutaneous, 1 gm dose of ceftriaxone (350 mg/mL solution administered at 2.5 mL/min over 1.14 minutes)
  Other Names: saline; normal saline; 0.9% sodium chloride injection
Drug: IV Ceftriaxone — single, intravenous infusion of 1 gm ceftriaxone (40 mg/mL solution administered at 0.83 mL/min over 30 minutes)
  Other Names: ceftriaxone

SUMMARY:
The objectives of this study are:

* to establish the safety of subcutaneous administration of ceftriaxone at different concentrations, with and without HYLENEX recombinant, and to determine the maximum tolerated concentration;
* and to establish the pharmacokinetic comparability of subcutaneous administration of ceftriaxone with HYLENEX recombinant to subcutaneous administration without HYLENEX recombinant and to IV administration.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18-65 years of age
* If female: non-lactating; non-pregnant; and incapable of becoming pregnant, or taking specific precautions to avoid becoming pregnant before and during study
* Normal clinical laboratory parameters
* Adequate venous access in both upper extremities
* Agreeing to refrain from smoking and from ingesting any alcohol or caffeine-containing products before and during the study
* Good health based on medical history, physical examination and laboratory tests
* Non-smoking; or smoking less than 10 cigarettes per day and willing to refrain from use of nicotine products before and during study

Exclusion Criteria:

* Received a cephalosporin within the 21 days prior to study or anticipated to receive non-study cephalosporin during study
* Pregnant or breast-feeding.
* Previously exposed to a hyaluronidase drug product
* Medical condition presenting unacceptable safety risk or likely to prevent completion of study
* Known hypersensitivity to hyaluronidase or any other ingredient in HYLENEX recombinant
* Contraindication to ceftriaxone, including known allergy to beta-lactam antibiotics
* Local condition precluding subcutaneous injection or injection site evaluation
* History of gastrointestinal disease (in particular colitis)
* Consumption of caffeine- or other methylxanthine-containing beverage within 24 hours before and/or during the PK sampling period
* Participation in study of any investigational drug or device within 30 days before this study
* Serum hemoglobin <12 g/dL.
* Blood donation or significant loss of blood within 56 days, or plasma donation within 7 days, prior to study
* Medical history/condition, screening physical examination finding or clinical laboratory result precluding safe participation in study, or which might adversely effect interpretation of study results
* History of drug or alcohol abuse within 2 years prior to study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-06; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George E Harb, MD, Study Director — Baxter Healthcare Corporation

REFERENCES:
- [Result] Harb G, Lebel F, Battikha J, Thackara JW. Safety and pharmacokinetics of subcutaneous ceftriaxone administered with or without recombinant human hyaluronidase (rHuPH20) versus intravenous ceftriaxone administration in adult volunteers. Curr Med Res Opin. 2010 Feb;26(2):279-88. doi: 10.1185/03007990903432900. PMID 19947907

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy volunteers recruited via subject-initiated telephone or internet contacts or visits to Phase I unit. Those considered potentially eligible were, after obtaining consent, screened in detail to determine eligibility against protocol eligibility criteria.
Groups:
- HYLENEX SC, Placebo SC, IV: subcutaneous HYLENEX and ceftriaxone as first intervention, subcutaneous placebo and ceftriaxone as second intervention, intravenous ceftriaxone as third intervention
- HYLENEX SC, IV, Placebo SC: subcutaneous HYLENEX and ceftriaxone as first intervention, intravenous ceftriaxone as second intervention, subcutaneous placebo and ceftriaxone as third intervention
- Placebo SC, HYLENEX SC, IV: subcutaneous placebo and ceftriaxone as first intervention, subcutaneous HYLENEX and ceftriaxone as second intervention, intravenous ceftriaxone as third intervention
- Placebo SC, IV, HYLENEX SC: subcutaneous placebo and ceftriaxone as first intervention, intravenous ceftriaxone as second intervention, subcutaneous HYLENEX and ceftriaxone as third intervention
- IV, HYLENEX SC, Placebo SC: intravenous ceftriaxone as first intervention, subcutaneous HYLENEX and ceftriaxone as second intervention, subcutaneous placebo and ceftriaxone as third intervention
- IV, Placebo SC, HYLENEX SC: intravenous ceftriaxone as first intervention, subcutaneous placebo and ceftriaxone as second intervention, subcutaneous HYLENEX and ceftriaxone as third intervention
Period: First Intervention
Arm/Group | HYLENEX SC, Placebo SC, IV | HYLENEX SC, IV, Placebo SC | Placebo SC, HYLENEX SC, IV | Placebo SC, IV, HYLENEX SC | IV, HYLENEX SC, Placebo SC | IV, Placebo SC, HYLENEX SC
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: First 7-Day Washout & Safety Follow-up
Arm/Group | HYLENEX SC, Placebo SC, IV | HYLENEX SC, IV, Placebo SC | Placebo SC, HYLENEX SC, IV | Placebo SC, IV, HYLENEX SC | IV, HYLENEX SC, Placebo SC | IV, Placebo SC, HYLENEX SC
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | HYLENEX SC, Placebo SC, IV | HYLENEX SC, IV, Placebo SC | Placebo SC, HYLENEX SC, IV | Placebo SC, IV, HYLENEX SC | IV, HYLENEX SC, Placebo SC | IV, Placebo SC, HYLENEX SC
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second 7-Day Washout & Safety Follow-up
Arm/Group | HYLENEX SC, Placebo SC, IV | HYLENEX SC, IV, Placebo SC | Placebo SC, HYLENEX SC, IV | Placebo SC, IV, HYLENEX SC | IV, HYLENEX SC, Placebo SC | IV, Placebo SC, HYLENEX SC
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention
Arm/Group | HYLENEX SC, Placebo SC, IV | HYLENEX SC, IV, Placebo SC | Placebo SC, HYLENEX SC, IV | Placebo SC, IV, HYLENEX SC | IV, HYLENEX SC, Placebo SC | IV, Placebo SC, HYLENEX SC
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 4 | 5 | 5 | 5 | 5 | 5
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Period: Final 7-Day Safety Follow-up
Arm/Group | HYLENEX SC, Placebo SC, IV | HYLENEX SC, IV, Placebo SC | Placebo SC, HYLENEX SC, IV | Placebo SC, IV, HYLENEX SC | IV, HYLENEX SC, Placebo SC | IV, Placebo SC, HYLENEX SC
Started | 4 | 5 | 5 | 5 | 5 | 5
Completed | 4 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HYLENEX SC, Placebo SC, IV | HYLENEX SC, IV, Placebo SC | Placebo SC, HYLENEX SC, IV | Placebo SC, IV, HYLENEX SC | IV, HYLENEX SC, Placebo SC | IV, Placebo SC, HYLENEX SC | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 5 | 5 | 5 | 5 | 30
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32.2 (10.6) | 37.6 (4.0) | 34.2 (11.5) | 34.8 (17.5) | 34.8 (11.0) | 33.2 (8.0) | 34.5 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 1 | 2 | 0 | 5
  Male | 4 | 5 | 4 | 4 | 3 | 5 | 25
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 5 | 5 | 5 | 5 | 30

OUTCOME MEASURES:

1. Secondary Outcome: Cmax
Description: Maximum measured plasma ceftriaxone concentration
Time Frame: at the time of the highest measured plasma ceftriaxone concentration
Population: Per protocol (excludes one participant that did not receive intravenous ceftriaxone intervention)
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- HYLENEX SC: All per-protocol participants administered subcutaneous hylenex and ceftriaxone
- Placebo SC: All per-protocol participants administered subcutaneous placebo and ceftriaxone
- Intravenous: All per-protocol participants administered intravenous ceftriaxone
Arm/Group | HYLENEX SC | Placebo SC | Intravenous
Number analyzed (Participants) | 29 | 29 | 29
µg/mL | 92.0 (15.1) | 82.2 (13.5) | 150 (19.9)
Statistical Analysis 1: Comparison: HYLENEX SC vs Placebo SC; Test type: Non-Inferiority or Equivalence — Bioequivalence = 90% confidence interval of least squares mean (LSM) within 80%-125%; Schuirmann two one-sided tests procedure; LSM ratio (natural log-transformed) = 111.79, 90% CI 2-sided [108.57 to 115.12] — HYLENEX SC/Placebo SC
Statistical Analysis 2: Comparison: HYLENEX SC vs Intravenous; Test type: Non-Inferiority or Equivalence — Bioequivalence = 90% confidence interval of least squares mean (LSM) within 80%-125%; Schuirmann two one-sided tests procedure; LSM ratio (natural log-transformed) = 60.81, 90% CI 2-sided [59.06 to 62.62] — HYLENEX SC/Intravenous
Statistical Analysis 3: Comparison: Placebo SC vs Intravenous; Test type: Non-Inferiority or Equivalence — Bioequivalence = 90% confidence interval of least squares mean (LSM) within 80%-125%; Schuirmann two one-sided tests procedure; LSM ratio (%; ln-transformed) = 54.40, 90% CI 2-sided [52.82 to 56.01] — Placebo SC/Intravenous

2. Secondary Outcome: Tmax
Description: Time to maximum measured plasma ceftriaxone concentration
Time Frame: from start of ceftriaxone administration until time of maximum measured plasma ceftriaxone concentration
Population: Per protocol (excludes one participant that did not receive intravenous ceftriaxone intervention)
Measure: Median (Full Range); unit: hr
Groups:
- Intravenous: All per-protocol participant administered intravenous ceftriaxone
Arm/Group | HYLENEX SC | Placebo SC | Intravenous
Number analyzed (Participants) | 29 | 29 | 29
hr | 2.02 [1.02 to 3.01] | 3.02 [1.52 to 4.04] | 0.502 [0.501 to 0.611]
Statistical Analysis 1: Comparison: HYLENEX SC vs Placebo SC; Test type: Superiority or Other; p < 0.01, Wilcoxon signed-rank test; Median Difference (Net) = -1.00, 90% CI 2-sided [-1.25 to -0.75] — HYLENEX SC minus Placebo SC
Statistical Analysis 2: Comparison: HYLENEX SC vs Intravenous; Test type: Superiority or Other; p < 0.01, Wilcoxon signed-rank test; Median Difference (Net) = 1.52, 90% CI 2-sided [1.27 to 1.71] — Placebo SC minus Intravenous
Statistical Analysis 3: Comparison: Placebo SC vs Intravenous; Test type: Superiority or Other; p < 0.01, Wilcoxon signed-rank test; Median Difference (Net) = 2.52, 90% CI 2-sided [2.26 to 2.76] — Placebo SC minus Intravenous

3. Primary Outcome: AUC0-t
Description: Area under the drug concentration-time curve from time zero to the time of the last measurable concentration (calculated by the linear trapezoidal method)
Time Frame: Start of ceftriaxone administration through time of last measureable plasma ceftriaxone concentration
Population: Per protocol (excludes one participant that did not receive intravenous ceftriaxone intervention)
Measure: Mean (Standard Deviation); unit: μg*hr/mL
Arm/Group | HYLENEX SC | Placebo SC | Intravenous
Number analyzed (Participants) | 29 | 29 | 29
μg*hr/mL | 1139.3 (200.30) | 1115.6 (180.55) | 1065.3 (176.07)
Statistical Analysis 1: Comparison: HYLENEX SC vs Placebo SC; Test type: Non-Inferiority or Equivalence — Bioequivalence = 90% confidence interval of least squares mean (LSM) within 80%-125%; Schuirmann two one-sided tests procedure; LSM ratio (%; ln-transformed) = 101.99, 90% CI 2-sided [98.95 to 105.12] — HYLENEX SC/Placebo SC
Statistical Analysis 2: Comparison: HYLENEX SC vs Intravenous; Test type: Non-Inferiority or Equivalence — Bioequivalence = 90% confidence interval of least squares mean (LSM) within 80%-125%; Schuirmann two one-sided tests procedure; LSM ratio (%; ln-transformed) = 106.79, 90% CI 2-sided [103.61 to 110.07] — HYLENEX SC/Intravenous
Statistical Analysis 3: Comparison: Placebo SC vs Intravenous; Test type: Non-Inferiority or Equivalence — Bioequivalence = 90% confidence interval of least squares mean (LSM) within 80%-125%; Schuirmann two one-sided tests procedure; LSM ratio (%; ln-transformed) = 104.71, 90% CI 2-sided [101.59 to 107.92] — Placebo SC/Intravenous

4. Primary Outcome: AUC0-inf
Description: Area under the drug concentration-time curve from time zero to infinity, calculated as AUC0-t + Ct/kel (Ct = time of last measurable concentration; kel = terminal elimination rate constant)
Time Frame: from the start of ceftriaxone administration to infinity
Population: Per protocol (excludes one participant that did not receive intravenous ceftriaxone intervention)
Measure: Mean (Standard Deviation); unit: µg*hr/mL
Arm/Group | HYLENEX SC | Placebo SC | Intravenous
Number analyzed (Participants) | 29 | 29 | 29
µg*hr/mL | 1162.6 (210.36) | 1141.3 (192.86) | 1085.8 (187.50)
Statistical Analysis 1: Comparison: HYLENEX SC vs Placebo SC; Test type: Non-Inferiority or Equivalence — Bioequivalence = 95% confidence interval of least squares mean (LSM) within 80%-125%; Schuirmann two one-sided tests procedure; LSM ratio (%; ln-transformed) = 101.76, 90% CI 2-sided [98.64 to 104.98] — HYLENEX SC/Placebo SC
Statistical Analysis 2: Comparison: HYLENEX SC vs Intravenous; Test type: Non-Inferiority or Equivalence — Bioequivalence = 90% confidence interval of least squares mean (LSM) within 80%-125%; Schuirmann two one-sided tests procedure; LSM ratio (%; ln-transformed) = 106.95, 90% CI 2-sided [103.67 to 110.33] — HYLENEX SC/Intravenous
Statistical Analysis 3: Comparison: Placebo SC vs Intravenous; Test type: Non-Inferiority or Equivalence — Bioequivalence = 90% confidence interval of least squares mean (LSM) within 80%-125%; Schuirmann two one-sided tests procedure; LSM ratio (%; ln-transformed) = 105.10, 90% CI 2-sided [101.87 to 108.42] — Placebo SC/Intravenous

ADVERSE EVENTS:
Time Frame: from time of start of intervention administration through 7 days after intervention administered
Description: Infusion site reaction assessments performed at baseline (shortly before study drug administration) and at 5, 30 and 45 minutes, and 1, 4, 6, 24, 36 and 48 hours after completion of study drug administration. Other adverse events were to be recorded whenever reported by the participant or observed by study staff.
Groups:
- HYLENEX SC: All participants administered subcutaneous HYLENEX and ceftriaxone
- Placebo SC: All participants administered subcutaneous placebo and ceftriaxone
- Intravenous: All participants administered intravenous ceftriaxone
Arm/Group | HYLENEX SC | Placebo SC | Intravenous
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 30/30 | 30/30 | 22/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HYLENEX SC (N=30) | Placebo SC (N=30) | Intravenous (N=29)
Infusion site anaesthesia (General disorders) | 4 | 1 | 0
Infusion site bruising (General disorders) | 2 | 4 | 6
Infusion site erythema (General disorders) | 18 | 15 | 4
Infusion site induration (General disorders) | 2 | 1 | 0
Infusion site pain (General disorders) | 30 | 30 | 9
Infusion site pruritus (General disorders) | 2 | 0 | 2
Infusion site reaction (General disorders) | 6 | 0 | 0 — Reported term = "muscle twitching"
Infusion site swelling (General disorders) | 5 | 28 | 1
Vessel puncture site bruise (General disorders) | 1 | 2 | 2 — Refers to site of placement of catheter for PK plasma sample collection, not study drug administration site
Headache (Nervous system disorders) | 2 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For this study, Baxter requires a review of any planned PI results communications (eg, for confidential information) up to 90 days prior to submission or communication. Baxter may request an additional delay of up to 60 days (eg, to allow for intellectual property protection).